CLINICAL TRIAL: NCT05504031
Title: Hybrid Revascularization Versus Coronary Artery Bypass Grafting in Patients With Multi-vessel Coronary Artery Disease. A Randomized Clinical Trial.
Brief Title: Hybrid Revascularization Versus Coronary Artery Bypass Grafting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); UMC Utrecht (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Christian Lildal Carranza, Chief Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hybrid-CABG Trial CPH
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Hybrid coronary revascularization; PCI; CABG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to Hybrid coronary revascularization or CABG
Who Masked: Investigator, Outcomes Assessor
Masking Description: We intend to blind all possible trial personal. Participants and care providers can not be blinded due to obvious scaring on the patient and the ward that is responsible for patient care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Group (Experimental): Revascularization in the form of a combined MIDCAB (LIMA-LAD graft trough a minimal invasive left anterior thoracotomy) and PCI (of all non-LAD stenoses)
  Interventions: Procedure: Hybrid coronary revascularization
- CABG Group (Active Comparator): Conventional CABG through a sternotomy
  Interventions: Procedure: Conventional revascularization

INTERVENTIONS:
Procedure: Hybrid coronary revascularization — Coronary revascularization is conducted as a combined MIDCAB (LIMA-LAD grafting through a minimally invasive anterior left thoracotomy) and PCI (of all non-LAD stenoses)
  Arms: Hybrid Group
Procedure: Conventional revascularization — Conventional revascularization with CABG of all significant stenoses through a sternotomy
  Arms: CABG Group

SUMMARY:
Coronary artery disease often necessitates complex interventions like coronary artery bypass surgery (CABG) or percutaneous coronary intervention (PCI) with stents. Hybrid coronary revascularization, a minimally invasive approach, integrates both methods for complete revascularization. This multicenter randomized trial involves 1200 patients, comparing hybrid coronary revascularization to CABG in a 1:1 ratio. Eligible participants have multi-vessel coronary disease and are referred for elective or sub-acute CABG. Inclusion criteria include age 18 or older, significant multi-vessel disease, and potential complete revascularization with both methods. Exclusion criteria include chronic kidney disease, pregnancy, contradiction to dual antiplatelet therapy, recent myocardial infarction, and acute revascularization. The hybrid group undergoes staged revascularization, combining minimally invasive grafting of the left interior mammary artery to the left anterior descending artery with PCI-stenting of remaining lesions. The control group undergoes conventional CABG with sternotomy. The primary outcome is a composite of all-cause mortality, myocardial infarction, stroke, or unplanned hospitalization, while secondary outcomes include periprocedural complications, cardiovascular mortality, hospital-free days within 90 days, angina frequency, and quality of life. Evaluation occurs 12 months after randomization. The trial commences in 2024, with inclusion expected to conclude in 5 years.

DETAILED DESCRIPTION:
Background

Cardiovascular diseases, mainly coronary artery disease (CAD), are the leading causes of death worldwide. CAD is characterized by the narrowing or blockage of blood flow in the coronary arteries often necessitating complex interventions like coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) with drug-eluting stents. The preferred revascularization strategy depends on several characteristics, one being the number of diseased vessels. Multivessel coronary artery disease (MVD) is defined as stenosis of at least two major coronary arteries.

Over the years, several large trials have concluded that CABG and PCI with newer-generation drug-eluting stents are both associated with improved survival rates compared to medical therapy.

CABG is still regarded as the gold standard for complex multivessel disease, with the cornerstone being the in-situ left internal mammary artery (LIMA) anastomosed to the left anterior descending artery (LAD).1 Current guidelines recommend CABG or PCI with equipoise in patients with one-vessel proximal LAD stenosis, two-vessel disease with proximal LAD stenosis, left main disease or three-vessel disease with lower complexity.2 The LIMA graft, with its excellent patency, has been shown to outperform PCI of the LAD and is in part responsible for the apparent success and survival benefit of CABG.3 However, saphenous vein grafts, the most common graft for non-LAD targets perform rather poorly, with graft failure ranging as high as 43%, 18 months after surgery.4 PCI with DES, especially with intravascular imaging, is documenting meagre failure rates and may consequently offer better results in non-LAD vessels than CABG with vein grafts does.5

Despite its survival benefits, the CABG comes at the cost of a full sternotomy, necessitating longer rehabilitation. Patients may prefer less invasive treatment options if these are feasible and have consistent long-term results. The minimally invasive coronary artery bypass (MIDCAB) procedure was developed as a less invasive method for revascularization. MIDCAB allows for the grafting of the anterior vessels through a small left anterior thoracotomy without the use of extracorporeal circulation. Thus, ensuring vital revascularization with a lesser trauma.

Complete revascularization has been established as the most important factor for survival. Recent data have showed comparable 10-year mortality in patients achieving this goal with either PCI or CABG.6

Hybrid coronary revascularization was developed to combine the best parts of the two revascularization techniques, consisting of a minimally invasive grafting of the LIMA to LAD, and PCI of all functionally significant non-LAD stenoses. Theoretically, patients may obtain the survival benefit from the LIMA-LAD graft, from a less invasive approach and avoidance of vein graft failures.

However, to this date, hybrid coronary revascularization is supported by very limited data. Only three small, randomized feasibility trials have been conducted, which all stated that the procedure is feasible but that larger randomized trials are necessary to determine if it is a suitable alternative to treating multivessel disease.7-9

Trial objective

The trial objective is to assess the beneficial and harmful effects of hybrid coronary revascularization versus coronary artery bypass graft surgery in patients with multivessel coronary artery disease.

Trial design

The trial investigaors will conduct a multicentre randomized superiority trial comparing hybrid coronary revascularization versus conventional CABG surgery in patients with multi-vessel coronary artery disease. Patients will be randomized 1:1 to hybrid coronary revascularization or CABG. The randomisation will be stratified according to clinical site and diabetes (yes/no).

Selection of participants

All patients with multi-vessel coronary disease referred for a CABG will be discussed during the heart team conference and considered for participation in the trial.

Inclusion criteria

* Written informed consent
* ≥ 18 years of age
* Functionally significant MVD, defined as ≥ 70% diameter stenosis by visual estimation or functionally significant stenosis (FFR < 0.80, non-hyperaemic index (iFR) < 0.89) in at least two of the major epicardial vessels or major side branches
* Patient history reviewed by both cardiac surgeon and cardiologist who in agreement find both CABG and hybrid revascularisation indicated and technically feasible with an expectation of complete revascularisation of all functionally significant stenoses in the LAD and at least one other coronary artery ≥ 2.5mm in diameter or left main bifurcation stenosis with functionally significant stenoses in both the LAD and left circumflex artery.

Exclusion criteria

* Chronic kidney disease with estimated glomerular filtration rate < 20 mL/min/kg
* Pregnancy
* Contraindications to the use of dual antiplatelet therapy
* STEMI within 1 month
* Indication for acute revascularization

Trial intervention

Experimental intervention:

Coronary revascularization will be conducted as a staged intervention. First, the MIDCAB will be conducted through a small left anterior thoracotomy, with endoscopic LIMA harvest and off-pump LIMA to LAD-grafting. Second, PCI with implantation of contemporary DES of all non-LAD lesions will be conducted within 4 weeks of the surgical procedure. Patients will receive dual antiplatelet therapy (DAPT) according to local routine and international guidelines.

A "reverse hybrid" with PCI preceding MIDCAB is also an option in patients with sub-acute coronary syndrome or CTO. Surgery will be conducted 3 months after PCI when it is safe to pause DAPT. PCI of CTO, guided by viability tests, may further be staged at up to 30 days after MIDCAB surgery.

Control intervention:

Coronary revascularization will be conducted as a conventional CABG, through a sternotomy, on- or off-pump with grafting of all target vessels, according to local best practice. All graft types are permitted and, therefore, surgeons decide their own specific graft strategy.

CABG, MIDCAB, and PCI are all standard procedures performed routinely at the hospitals. Therefore, there is no expected increased risk for trial participants no matter which group they are randomized to.

The statistical analysis will adhere to the intention-to-treat principle, meaning that participants will be analyzed based on their originally assigned groups even if they undergo a crossover to other interventions.

Outcome measures

Primary outcome

• A composite outcome of either all-cause mortality, a diagnosis of myocardial infarction, a diagnosis of stroke, or any unplanned hospitalization at 12 months postoperatively.

Secondary outcomes

* Periprocedural complications defined as periprocedural myocardial infarction, stroke, unplanned re-intervention, BARC 3-5 bleeding complications10, or surgical wound infection.
* Cardiovascular mortality
* Hospital free days within 90 days after randomization
* Angina frequency using the Seattle Angina Questionnaire11
* Health-related quality of life using EQ-5D12

Exploratory outcomes

* Serious adverse events (dichotomous). We will use the International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use-Good Clinical Practice (ICH-GCP) definition of a serious adverse event, which is any untoward medical occurrence that resulted in death, was life-threatening, required hospitalisation or prolonging of existing hospitalisation and resulted in persistent or significant disability or jeopardised the participant.
* Major Adverse Kidney Events to 30 days (MAKE30), defined as either death, new renal replacement therapy, or persistent renal dysfunction (creatinine at discharge or day 30 ≥ 200% of the baseline serum creatinine value)
* Post-pericardiotomy syndrome (diagnosed by two of the following being present: fever without alternative cause, pleuritic chest pain, friction rub on auscultation and evidence of new or worsening pericardial or pleural effusion)
* Postoperative pain
* Need for reoperation
* Prolonged intubation (> 48 hours)
* Acute kidney injury within 48 hours, defined by the KDIGO criteria
* Biomarkers during hospital stay (e.g. CK-MB, troponins, creatinine, haemoglobin)
* Length of stay
* Urgent revascularization or myocardial infarction
* Admission for new onset of heart failure
* Completeness of index revascularization
* Target vessel failure
* Target vessel revascularization
* Any repeat revascularization
* Definite stent thrombosis
* Atrial fibrillation (AF) within 3 months of revascularization (AF will be handled according to local practice)
* Sternal wound infections - superficial and deep
* Sternal wound dehiscence
* New York Heart Association (NYHA) class
* Healthcare costs
* Major arrhythmia within 30 days (supraventricular tachycardia requiring cardioversion, ventricular tachycardia or fibrillation requiring treatment, or bradyarrhythmia requiring temporary or permanent pacemaker)
* Graft failure assessed on cardiac computed tomography (CT) at 1 year (if the procedure is conducted)

Sample size and power estimation

Provided that the incidence of all-cause mortality, a diagnosis of myocardial infarction, a diagnosis of stroke, or hospitalization in the control group is equal to 55%, an absolute risk reduction of 10% (corresponding to a relative risk reduction of 18.2%), α=0.05, beta=0.10 (giving a power of 90%) we will need 524 participants in the intervention and in the control group. Notably, a 10% absolute risk reduction corresponds to an incidence of either all-cause mortality, a diagnosis of myocardial infarction, a diagnosis of stroke, or hospitalization equal to 45% in the experimental intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥ 18 years of age
* Functionally significant MVD, defined as ≥ 70% diameter stenosis by visual estimation or functionally significant stenosis (FFR < 0.80, non-hyperaemic index (iFR) < 0.89) in at least two of the major epicardial vessels or major side branches
* Patient history reviewed by both cardiac surgeon and cardiologist who in agreement find both CABG and hybrid revascularisation indicated and technically feasible with an expectation of complete revascularisation of all functionally significant stenoses in the LAD and at least one other coronary artery ≥ 2.5mm in diameter or left main bifurcation stenosis with functionally significant stenoses in both the LAD and left circumflex artery.

Exclusion Criteria:

* Chronic kidney disease with estimated glomerular filtration rate < 20 mL/min/kg
* Pregnancy
* Left main stenosis without additional functionally significant stenoses in both the LAD and the LCX
* Contraindications to the use of dual antiplatelet therapy
* STEMI within 1 month
* Indication for acute revascularization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
A composite outcome of either all-cause mortality, a diagnosis of spontaneous myocardial infarction, a diagnosis of stroke, or any unplanned hospitalization | 12 months after randomization
  A composite outcome of either all-cause mortality, a diagnosis of spontaneous myocardial infarction, a diagnosis of stroke, or any unplanned hospitalization

SECONDARY OUTCOMES:
Angina symptoms | 12 months after randomization
  Angina symptoms measured using Seattle Angina Questionnaire
Health related quality of life | 12 months after randomization
  Health related quality of life using EQ-5D
Hospital free days | 90 days after randomization
  Hospital free days
Procedural complications | 12 months after randomization
  Procedural complications defined as periprocedural myocardial infarction, unplanned re-intervention, stroke, BARC 3-5 bleeding complications or sternal wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Christian Carranza, MD, E-MBA, Study Director — Department of Cardiothoracic Surgery, Copenhagen University Hospital, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We plan to make all data publicly available in peer-review papers, after the trial has been finalized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the trial
Access Criteria: In peer-review papers